CLINICAL TRIAL: NCT04998435
Title: Ultrasound-Guided Paravertebral Block Versus Erector Spinae Plain Block For Perioperative Analgesia In Adults Undergoing Percutaneous Nephrolithotomy: A Randomized Clinical Trial
Brief Title: Paravertebral Block Versus Erector Spinae Plain Block In Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nazmy Edward Seif (Other)
Responsible Party: Sponsor-Investigator, Nazmy Edward Seif, Clinical Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PVBVESPBPCNL
Record Dates: First submitted 2021-07-27; First posted 2021-08-10 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Renal Stone; Nephrolithiasis; Analgesia; Anesthesia
Keywords: Erector spinae plain block; Paravertebral block; Ultrasound-guided; Percutaneous nephrolithotomy; Analgesia
MeSH Terms: conditions — Nephrolithiasis; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB group (Active Comparator): Erector Spinae Plain Block
  Interventions: Procedure: Erector Spinae Plain Block
- PV group (Active Comparator): Paravertebral Block
  Interventions: Procedure: Paravertebral Block

INTERVENTIONS:
Procedure: Erector Spinae Plain Block — Using aseptic technique, ultrasound-guided ESPB will be performed with the patient in sitting position. The spinous process of the vertebra and a point 3 cm lateral to it will be marked before performing the block. The needle will be inserted and advanced under sono-visualization to contact the transverse process of the vertebra. After negative aspiration, LA will be deposited into the fascial plane deep to erector spinae muscle.
  30 ml of Bupivacaine 0.25% will be used as LA, injected using a 22-gauge spinal needle at the level of T10 which will be identified by counting 3 spinous processes below T7 which is at the level of the inferior angle of the scapula and also rechecked by counting down from C7.
  Patients will then receive general anesthesia. All patients will receive paracetamol (1gm/8hrs IV) as a regular analgesia. IV morphine (0.02mg/kg) will be given as a rescue analgesia if the Visual Analogue Scale for pain is ≥ 4.
  Arms: ESPB group
Procedure: Paravertebral Block — Using sterile technique, ultrasound scanning of thoracic paravertebral space will be done in sitting position. The transverse process will be identified as hyperechoic structure while pleura will be identified as a mobile hypoechoic structure. The needle will be inserted cranio-caudal and advanced under sono-visualization to the identified thoracic paravertebral space. After negative aspiration, LA will be deposited displacing the pleura.
  30 ml of Bupivacaine 0.25% will be used as LA, injected using a 22-gauge spinal needle at the level of T10 which will be identified by counting 3 spinous processes below T7 which is at the level of the inferior angle of the scapula and also rechecked by counting down from C7.
  Patients will then receive general anesthesia. All patients will receive paracetamol (1gm/8hrs IV) as a regular analgesia. IV morphine (0.02mg/kg) will be given as a rescue analgesia if the Visual Analogue Scale for pain is ≥ 4.
  Arms: PV group

SUMMARY:
Nowadays, Percutaneous Nephrolithotomy (PCNL) has been the surgical procedure of choice for renal stones larger than 2cm or staghorn stones. Yet, the associated postoperative pain is a major drawback. The regional anesthetic management of pain in PCNL operation has been of great concern. The introduction of ultrasound guided erector spinae plane block and paravertebral plane block has been under great focus regarding the efficacy of postoperative pain management. Paravertebral plane block (PVB) is a regional nerve block technique that depends on local anesthetic injection adjacent to the vertebra to block spinal nerve roots in a dermatomal distribution. Erector spinae plane block (ESPB) is a newer regional anesthesia technique that depends on injecting local anesthetic (LA) in a plane between the transverse process and erector spinae muscle. The LA diffuses into the paravertebral space and spreads on both rami (dorsal and ventral) of spinal nerves through spaces between adjoining vertebrae.

The aim of this study is to compare the effect of ultrasound guided Paravertebral blockade versus Erector spinae blockade on postoperative opioid use as well as postoperative pain control in patients undergoing unilateral PCNL.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II.
* Patients undergoing unilateral percutaneous nephrolithotomy (PCNL) surgery under general anesthesia.

Exclusion Criteria:

* Patient refusal.
* Uncooperative patients.
* Allergy to local anesthetics.
* Infection or anatomical abnormality at injection site.
* Coagulopathy.
* Bilateral PCNL.
* Spinal anesthesia or any other regional anesthesia.
* Block failure: the block will be considered a failed block if the patient requires more than two doses of rescue analgesia in the first hour postoperatively.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Morphine consumption. | 24 hours
  Total dose of Morphine (measured in mg) given intra-venously to the patient post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Atef K Salama, MD, Study Director — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University.; Nazmy S Michael, MD, Study Chair — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University.
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided